CLINICAL TRIAL: NCT02725723
Title: Thermographic Images as an Objective Method for Assessing the Efficacy of Steroidal Epidural Injections
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Chief Executive Officer, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-16-SB-0650-15-CTIL
Record Dates: First submitted 2016-03-21; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subject after epidural injection (Experimental): Subjects are patients from the clinic who have been diagnosed with Lumbar spinal stenosis and determined eligible for receiving steroidal epidural injection for pain management
  Interventions: Device: Therm-AppTM TH, thermographic camera; Drug: epidural injection

INTERVENTIONS:
Device: Therm-AppTM TH, thermographic camera
Drug: epidural injection

SUMMARY:
Spinal stenosis is a prevalent diagnosis, which is handled in a heterogeneous manner by clinicians. Moreover, when using steroidal epidural injections, successful treatment is currently defined as the satisfaction of the patient from the treatments, a subjective and non-quantifiable indicator.

In this experiment, the investigators aim to evaluate thermographic images as an objective method for assessing the efficacy of steroidal epidural injections, the most common invasive treatment for pain associated with spinal stenosis

ELIGIBILITY:
Inclusion Criteria:

* Signed a valid, IRB/EC-approved informed consent form
* 18 years of age or older when written informed consent is obtained
* Diagnosis of spinal stenosis by MRI or CT imaging

Exclusion Criteria:

* Sensitivity to local anesthetics
* Skin infection at the site of needle insertion
* Had evidence of a peripheral neuropathy
* Had clinical signs of peripheral vascular disease
* Patient is pregnant
* Clinical diagnosis of blood clotting disorder
* Tumor or infection at spine as demonstrate at MRI Unbalanced Cardiac Insufficiency, hypertension & Diabetes cataract Stomach Ulcer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Changes in Ts (Skin Temperature) will be determined at image taken by Therm-AppTM TH camera at the same region | Baseline and 30 min

SECONDARY OUTCOMES:
Change in Pain Intensity by a 0 - 10 numerical rating scale (NRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine". | Baseline, 1 month, 3 months

IPD SHARING:
Plan to Share IPD: No